CLINICAL TRIAL: NCT04352166
Title: Randomized Controlled Trial of Extended-Release Buprenorphine vs. Sublingual Buprenorphine for the Treatment of Opioid Use Disorder Patients Using Fentanyl
Brief Title: Extended-Release Buprenorphine vs. Sublingual Buprenorphine for the Treatment of Opioid Use Disorder
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: U.S. Department of Health and Human Services OHRP issued an FWA restriction on NYSPI research that included a pause of human subjects research as of June 23, 2023. This study will resume recruitment after OHRP has approved the resumption of research.
Sponsor: Frances R Levin (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Frances R Levin, Research Psychiatrist, New York State Psychiatric Institute
Organization: New York State Psychiatric Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7963; R21DA049037 (NIH)
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Opioid-use Disorder
Keywords: opioid use disorder; fentanyl; treatment; Sublocade
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Sublocade; Buprenorphine

STUDY DESIGN:
Intervention Model Description: Two arm, randomized (1:1 allotment), open-label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- extended-release buprenorphine (BXR) (Experimental): Three extended-release buprenorphine (BXR) injections to be administered roughly 28 days apart. The first and second injection will be 300 mg and the third will be 100 mg.
  Interventions: Drug: extended-release buprenorphine (BXR)
- sublingual buprenorphine (BSL) (Active Comparator): sublingual buprenorphine (BSL) up to 24 mg will be administered once daily for 12 weeks or length of study participation.
  Interventions: Drug: sublingual buprenorphine (BSL)

INTERVENTIONS:
Drug: extended-release buprenorphine (BXR) — Three monthly injections will be provided during the course of the 12 week trial.
  Other Names: Sublocade
  Arms: extended-release buprenorphine (BXR)
Drug: sublingual buprenorphine (BSL) — On a weekly basis patients will be provided with sublingual buprenorphine to take up to 24 mg daily.
  Other Names: buprenorphine
  Arms: sublingual buprenorphine (BSL)

SUMMARY:
The study is 12-week, randomized, open-label study comparing injectable extended-release buprenorphine (Sublocade) to standard therapy (sublingual buprenorphine), to see if Sublocade will be more helpful in treating opiate use for individuals testing positive for fentanyl and related high potency drugs (HPSO). Those receiving Sublocade will have it administered monthly and dosing will be according to the FDA prescribing instructions of 300mg for the first and second dose and 100mg for the third. Individuals receiving sublingual buprenorphine will receive standard dosing for the entire treatment trial. Participants will be asked to attend the clinic for the first 4 days during week 1 and twice weekly for the remainder of the trial.

DETAILED DESCRIPTION:
Outpatients seeking treatment for Opioid Use Disorder (OUD) will be screened, and those eligible and consenting will be randomized (n=40) to either buprenorphine extended-release (BXR, Sublocade) or sublingual buprenorphine (BSL). Randomization will occur in a 1:1 ratio immediately prior to starting the induction process. The primary hypothesis is that BXR treatment will significantly reduce opioid use as compared to BSL. This is a 12 week outpatient trial during which participants will be asked to come into the clinic for the first 4 days of week 1 and then twice weekly there after.

For buprenorphine to be safely administered, participants must be in withdrawal from opioids. Individuals will be instructed to abstain from opioids starting at consent and will usually begin buprenorphine medication within 24 hours of consent. Because HPSO use may lead to a delayed onset of opioid withdrawal syndrome, the first day that buprenorphine is administered may not be up to three days after a participants last opioid use. Whichever day the first dose of BSL is administered will be considered the first day of the induction.

BXR Injection group. There are two dosing schemes for the BXR induction as outlined below:

a) If on any day of the buprenorphine induction a participant demonstrates a high tolerance to buprenorphine by tolerating 24 mg buprenorphine SL in one day, BXR 300 mg may be administered on that study day. This includes participants who on the first day of SL buprenorphine administration tolerate 24 mg. b) If a patient is able to tolerate 16 mg of buprenorphine SL for 2 consecutive days of the induction, BXR 300 mg will be given on the second consecutive day of receiving buprenorphine SL 16 mg. The second injection of BXR 300 mg will be administered approximately 28 days later. The third BXR injection will occur approximately 28 days subsequent to the second injection at a dose of 100 mg.

Maintenance BSL treatment group: Once a participant is able to be stabilized on 16 mg to 24 mg per day during induction they will continue to receive buprenorphine in doses up to 24 mg administered once daily. Dose adjustments for craving/withdrawal/adverse effects will be made by the research psychiatrist. Medication will be dispensed on a weekly basis.

For both study arms participants will be given comfort medications to help manage their withdrawal for the first two weeks of the treatment study as needed. Comfort medications prescribed will be clonidine, clonazepam, prochlorperazine, and zolpidem.

If a participant is not in adequate withdrawal to be able to start sublingual buprenorphine (i.e., they continue to use once enrolled), they will have up to 10 days to initiate the induction for either arm of the study. If a participant is unable to start sublingual buprenorphine within 10 days of signing consent they will be considered an induction fail and will be provided referrals for other treatment options noted in the discontinuation section of the protocol.

At each visit, patients will be seen by the Research Nurse and Research Assistant for assessment of vital signs, side effects and adverse events, collection of urine for toxicology, and research assessments. The research psychiatrist will conduct weekly assessments of the psychiatric and medical status of the study participants. All participants will have a manual-guided supportive behavioral treatment session with the research psychiatrist each week. This psychosocial intervention facilitates compliance with study medication and other study procedures, promotes abstinence from opioids and other substances.

Post-study Assessments and Clinical Follow up: At week 12 (or earlier if the patient is discontinued from the study for clinical reasons or drops out) participants will be provided with clinical referrals for continuation of treatment. Post-study participants will be seen weekly for up to 4 weeks while continuing treatment with buprenorphine. Referrals will be arranged during this period for patients to continue buprenorphine or other appropriate treatment at community-based treatment programs.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the age of 18-65
* Voluntarily seeking treatment for opioid use
* Meets current DSM-5 criteria for Opioid Use Disorder as a primary diagnosis, with at least moderate severity
* Test positive for high potent synthetic opioids (HPSO) use
* Able to provide informed consent and comply with study procedures

Exclusion Criteria:

* Meets DSM-5 criteria for substance use disorder other than opioid as the primary diagnosis
* Having a comorbid psychiatric diagnosis that might interfere with participation or make participation hazardous, such as an active psychotic disorder or current suicide risk
* Methadone maintenance treatment within the past 30 days
* Buprenorphine maintenance treatment within the past 30 days
* Known history of allergy, intolerance, or hypersensitivity to candidate medication (buprenorphine)
* Pregnancy, lactation, or failure to use adequate contraceptive methods in female patients; male participants are required to use adequate forms of birth control as the exposure to sublocade on sperm and subsequent fetal development are not known
* Unstable medical conditions, which might make participation hazardous such as uncontrolled hypertension (blood pressure >150/100), acute hepatitis, uncontrolled diabetes, or elevated liver function tests (AST and ALT >3 times the upper limit of normal
* Legally mandated to substance use disorder treatment
* Current physiological dependence on alcohol or sedative-hypnotics that would require a medically supervised detoxification-other substance use diagnoses are not exclusionary
* Individuals, who in the clinicians judgment, have a history of failed trial of buprenorphine or sublocade (e.g., history of severe opioid intoxication or overdoses despite adequate adherence to buprenorphine or sublocade), or other features of the history strongly suggest the patient is not a good candidate for outpatient treatment with buprenorphine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Days of opioid use per week | up to 12 weeks
  Days of opioid use per week as measured by the timeline follow-back method and confirmed by urine toxicology.

CONTACTS AND LOCATIONS:
Overall Officials: frances r levin, md, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Nyspi-Stars, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results published in this report (after de-identification) (text, tables, figures)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning twelve months and ending 5 years after article publication
Access Criteria: to researcher who provides a methodologically sound proposal to achieve aims in approved proposal